CLINICAL TRIAL: NCT01071265
Title: Remote Ischemic Preconditioning in Cardiac Surgery: a Pilot Randomized Controlled Trial
Brief Title: Remote Ischemic Preconditioning in Cardiac Surgery Trial
Acronym: Remote IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-536; NIF-09223 (Other Grant/Funding Number: Hamilton Health Sciences New Investigator Fund); CANNeCTIN Funding (Other Grant/Funding Number: Canadian Network and Centre for Trials Internationally)
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Cardiac Surgery
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham RIPC (Placebo Comparator): Inflation of thigh pneumatic tourniquet to <15 mmHg
  Interventions: Procedure: Sham
- Active RIPC (Active Comparator): 300 mmHg inflation of thigh pneumatic tourniquet for three cycles of 5 minutes each with 5 minutes of no inflation between cycles.
  Interventions: Procedure: Remote Ischemic Preconditioning

INTERVENTIONS:
Procedure: Remote Ischemic Preconditioning — Occlusion of leg blood flow using a pneumatic tourniquet on the thigh. Tourniquets are inflated to 300 mmHg for 5 minutes followed by deflation for 5 minutes then repeated for a total of 3 inflations.
  Arms: Active RIPC
Procedure: Sham — Sham procedure. A pneumatic tourniquet is placed on an upper arm and/or thigh but not inflated.
  Arms: Sham RIPC

SUMMARY:
Main Research Questions:

1. Is a large trial of patients undergoing heart surgery comparing a simple procedure of temporarily stopping blood flow to the leg with a blood pressure cuff (called remote ischemic preconditioning) to a sham procedure possible?
2. Does the remote ischemic preconditioning procedure before heart surgery help protect the heart and kidneys?

What is Being Studied:

A simple procedure known as remote ischemic preconditioning. The procedure is performed by inflating a pressurized cuff the thigh to temporarily stop blood flow to the arm or leg. This procedure causes the body to have a stress response that, at the cellular level, may protect major organs like the heart and kidney from the damage caused to them by the much larger stress of cardiac surgery. Reducing this damage may improve patient's recovery after surgery and help them live longer.

Why is this study important?:

This research is important because up to 1 in every 20 patients that undergo heart surgery die before even leaving hospital. Preventing heart and kidney damage at the time of surgery with remote ischemic preconditioning may reduce patient deaths.

DETAILED DESCRIPTION:
Annually, 2 million patients worldwide undergo heart surgery. Although this procedure can prolong life, 1 in 20 patients will not survive their hospital stay. Acute heart and kidney injuries are important causes of death after heart surgery. Remote ischemic preconditioning (RIPC) is a promising and simple therapy that may simultaneously reduce heart and kidney damage. RIPC involves the inflation of a tourniquet or blood pressure cuff on a limb to briefly stop blood flow to that limb. This period of no blood flow activates the body's own protective systems and releases protective chemicals into the blood that also protect the heart and kidneys. RIPC is a particularly attractive potential treatment because it may protect several organs at once, it has no known adverse effects and costs almost nothing. RIPC could therefore very easily be used globally to improve outcomes for all patients undergoing heart surgery. Although RIPC appears very promising in several small studies using different RIPC regimens there are no studies large enough to definitively evaluate whether RIPC improves patient important outcomes (e.g. survival, kidney failure, major heart attack, or stroke). Before performing a large trial to determine whether RIPC is effective, we must demonstrate that such a trial is feasible. We will determine the recruitment rate and adequacy of follow-up in an international group of centres to ensure that an adequately powered trial of RIPC compared to a sham procedure is possible. Further, we will ensure that our RIPC regimen is consistent with other trials in terms of effects on cardiac and kidney injury. This pilot trial will enroll 250 patients and randomize half to RIPC and half to a sham procedure. We call this trial the Remote IscheMia Preconditioning in cArdiaC surgery Trial (Remote IMPACT).

ELIGIBILITY:
Inclusion Criteria:

* undergoing cardiac surgery
* at least 18 years old
* EuroSCORE >= 6

Exclusion Criteria:

* requiring intra-aortic balloon pump support prior to surgery
* unable to provide informed consent or decline to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2011-03; Primary Completion 2012-05 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Peak CK-MB within 24 hours after surgery | 24 hours
  Peak CK-MB within 24 hours after surgery

SECONDARY OUTCOMES:
Change in serum creatinine | within 4 days after surgery
All-cause mortality | 6 months after surgery
Need for Dialysis | 6 months after surgery
Length of hospital stay | Discharge from hospital after surgery
Length of stay in the intensive care unit | Discharge from hospital after surgery
Incidence of pneumonia | 30 days after surgery
Incidence of stroke | 6 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Michael Walsh, MD MSc, Principal Investigator — McMaster University; PJ Devereaux, MD PhD, Principal Investigator — McMaster University
Locations (7):
- United States (2):
  - Maine Medical Centre, Portland, Maine
  - Wake Forest, Winston-Salem, North Carolina
- Canada (5):
  - University of Calgary, Calgary, Alberta
  - Maritime Heart Centre, Halifax, Nova Scotia
  - McMaster University, Hamilton, Ontario
  - Lawson Health Research Institute, London, Ontario
  - Sunnybrook Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Walsh M, Whitlock R, Garg AX, Legare JF, Duncan AE, Zimmerman R, Miller S, Fremes S, Kieser T, Karthikeyan G, Chan M, Ho A, Nasr V, Vincent J, Ali I, Lavi R, Sessler DI, Kramer R, Gardner J, Syed S, VanHelder T, Guyatt G, Rao-Melacini P, Thabane L, Devereaux PJ; Remote IMPACT Investigators. Effects of remote ischemic preconditioning in high-risk patients undergoing cardiac surgery (Remote IMPACT): a randomized controlled trial. CMAJ. 2016 Mar 15;188(5):329-336. doi: 10.1503/cmaj.150632. Epub 2015 Dec 14. PMID 26668200